CLINICAL TRIAL: NCT04441684
Title: Study of the Seroprevalence of SARS-CoV-2 in Hospital Staff in Strasbourg University Hospital, Strasbourg, France
Brief Title: Seroprevalence of SARS-CoV-2 in Strasbourg University Hospital, Strasbourg, France (COVID-19)
Acronym: SeroCoV-HUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 7782
Record Dates: First submitted 2020-05-20; First posted 2020-06-22 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: SARS-CoV-2 Serological Status; SARS-CoV-2 Seroprevalence
Keywords: COVID-19; SARS-CoV-2; Humoral response; T-cell response
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection; Serologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PCR+ group (Experimental): This group includes any symptomatic person with a positive COVID result, with a RT-PCR test carried out at least 10 days before inclusion.
  Interventions: Diagnostic Test: Blood sample for serological test
- PCR- group (Experimental): This group includes any symptomatic person with a negative RT-PCR COVID 19 test carried out at least 10 days before inclusion.
  Interventions: Diagnostic Test: Blood sample for serological test
- No PCR (Experimental): This group includes any person, for which no COVID 19 RT- PCR testing was performed.
  Interventions: Diagnostic Test: Blood sample for serological test

INTERVENTIONS:
Diagnostic Test: Blood sample for serological test — Serology tests:
  * By LFA-ICT: BIOSYNEX COVID-19 BSS reference SW40005, BIOSYNEX SWISS SA, Fribourg, Switzerland
  * ELISA: EDI™ Novel Coronavirus COVID-19 ELISA IgG Kit, Epitope Diagnostics, Inc., San Diego, USA
  Confirmation test by seroneutralization tests developed at the Strasbourg Virology laboratory on whole virus (analyzes performed in a biosafety level 3 laboratory) and by the viral pseudoparticles system, will be performed.

SUMMARY:
COVID-19 is a new emerging disease caused by infection with the SARS-CoV-2 coronavirus, with no specific therapeutic options.

Since the end of February 2020, the Strasbourg University Hospital (HUS) had faced a sudden increase of patients with COVID-19 resulted from a SARS-CoV-2 superspreading event (religious meeting). Infected individuals went to regional hospitals, and this led to a cluster of infected healthcare workers at the Strasbourg University Hospitals from the first week of March. To date, several hundred Strasbourg hospital workers have presented a SARS-CoV-2 infection confirmed by the RT-PCR test from a nasopharyngeal sample. Most of them developed a mild form of COVID-19.

It is important to understand how far the infection has spread in the hospital staff, and to which extent the individuals who have been infected develop antibodies against SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

* Any person, male or female, over 18 years of age at the time of signing the consent
* Any person affiliated to a social health insurance scheme
* Any person able to understand the objectives and risks related to research and to give an informed, dated and signed consent
* Any person who is part of HUS staff and working at HUS at the time of the pandemic, including residents affiliated with HUS and assigned to general hospitals in the region
* Any symptomatic person with a positive COVID result (PCR + group) or negative (PCR- group) with a RT-PCR test carried out at least 10 days before inclusion, or any person, for which no COVID PCR was performed (group " No PCR")

Exclusion Criteria:

* Person in exclusion period (determined by a previous or ongoing study),
* Inability to give clear information (person in an emergency, difficulty understanding the subject, etc.)
* Person under safeguard of justice
* Person under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1466 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Presence of specific SARS-CoV2 antibodies in the serum in the 3 groups of subjects studied, at the inclusion visit (D0). | inclusion visit (Day 0).
  Presence of specific SARS-CoV2 antibodies in the serum in the 3 groups of subjects studied, at the inclusion visit (D0).

SECONDARY OUTCOMES:
Detection and titration of neutralizing antibodies anti-SARS-CoV-2 | At Day 0 and each follow-up visits i.e. at Month 3 (Day 0+3 months), Month 6 (Day 0+6 months) and Month 12 (Day 0+12 months).
Kinetics of antibodies and their persistence over a period of 1 year | At Day 0 and each follow-up visits i.e. at Month 3 (Day 0+3 months), Month 6 (Day 0+6 months) and Month 12 (Day 0+12 months).
Number of asymptomatic subjects in the PCR - and -PCR groups | At Day 0 and each follow-up visits i.e. at Month 3 (Day 0+3 months), Month 6 (Day 0+6 months) and Month 12 (Day 0+12 months).
Number of people with positive Sars-CoV-2 serology | At Day 0 and each follow-up visits i.e. at Month 3 (Day 0+3 months), Month 6 (Day 0+6 months) and Month 12 (Day 0+12 months).
Questionnaire (Type of health care personnel, Contact history, medical operation and respect of hygiene standards) | At Day 0 and each follow-up visits i.e. at Month 3 (Day 0+3 months), Month 6 (Day 0+6 months) and Month 12 (Day 0+12 months).

OTHER OUTCOMES:
Analysis of the T cell response by the ELISPOT technique | At one of the follow up visit : Month 3 (Day 0+3 months), Month 6 (Day 0+6 months) or Month 12 (Day 0+12 months).
B cell repertoire sequencing | At one of the follow up visit : Month 3 (Day 0+3 months), Month 6 (Day 0+6 months) or Month 12 (Day 0+12 months).
Sequencing of cellular SARS-CoV2 receptors | At one of the follow up visit : Month 3 (Day 0+3 months), Month 6 (Day 0+6 months) or Month 12 (Day 0+12 months).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg - Centre d'Investigation Clinique - Nouvel Hôpital Civil et Hautepierre, Strasbourg, France

REFERENCES:
- [Background] Garcia L, Woudenberg T, Rosado J, Dyer AH, Donnadieu F, Planas D, Bruel T, Schwartz O, Prazuck T, Velay A, Fafi-Kremer S, Batten I, Reddy C, Connolly E, McElheron M, Kennelly SP, Bourke NM, White MT, Pelleau S. Kinetics of the SARS-CoV-2 Antibody Avidity Response Following Infection and Vaccination. Viruses. 2022 Jul 8;14(7):1491. doi: 10.3390/v14071491. PMID 35891471
- [Result] Gallais F, Gantner P, Bruel T, Velay A, Planas D, Wendling MJ, Bayer S, Solis M, Laugel E, Reix N, Schneider A, Glady L, Panaget B, Collongues N, Partisani M, Lessinger JM, Fontanet A, Rey D, Hansmann Y, Kling-Pillitteri L, Schwartz O, De Seze J, Meyer N, Gonzalez M, Schmidt-Mutter C, Fafi-Kremer S. Evolution of antibody responses up to 13 months after SARS-CoV-2 infection and risk of reinfection. EBioMedicine. 2021 Sep;71:103561. doi: 10.1016/j.ebiom.2021.103561. Epub 2021 Aug 27. PMID 34455390